CLINICAL TRIAL: NCT05358587
Title: Comparison of the Perioperative Analgesic Efficacy of PENG Block Applications With Two Different Volumes in Patients Undergoing Hip Surgery
Brief Title: PENG Block With Two Diffirent Volume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, Gamze Ertas, anesthesiologist, Samsun University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PENG_55
Record Dates: First submitted 2022-04-20; First posted 2022-05-03 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Pain, Acute; Postoperative Pain; Hip Fractures
MeSH Terms: conditions — Acute Pain; Pain, Postoperative; Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG (20 mL) (Experimental): In this group, US guided PENG block will be performed with 20 ml of Bupivacaine solution (0.25 %)
  Interventions: Other: Ultrasound guided PENG block with 20 mL Local Anesthetic solution
- PENG (30 mL) (Experimental): In this group, US guided PENG block will be performed with 30 ml of Bupivacaine solution (0.25 %)
  Interventions: Other: Ultrasound guided PENG block with 30 mL Local Anesthetic solution

INTERVENTIONS:
Other: Ultrasound guided PENG block with 20 mL Local Anesthetic solution — In this group, US guided PENG block will be performed with 20 ml of Bupivacaine solution (0.25 %). Block will be performed 30 minutes before spinal anesthesia.
  Arms: PENG (20 mL)
Other: Ultrasound guided PENG block with 30 mL Local Anesthetic solution — In this group, US guided PENG block will be performed with 20 ml of Bupivacaine solution (0.25 %). Block will be performed 30 minutes before spinal anesthesia.
  Arms: PENG (30 mL)

SUMMARY:
Hip fractures are morbid conditions, especially in elderly patients, and their treatment is usually surgical. Pericapsular nerve group block is a newly defined block and targets the hip capsule. The aim of this study is to investigate and compare the perioperative analgesic efficacy of PENG blocks applied in two different volumes in patients undergoing hip fracture surgery under spinal anesthesia.

DETAILED DESCRIPTION:
Hip fractures are morbid conditions, especially in elderly patients, and their treatment is usually surgical. Pericapsular nerve group block is a newly defined block and targets the hip capsule. The aim of this study is to investigate and compare the perioperative analgesic efficacy of PENG blocks applied in two different volumes in patients undergoing hip fracture surgery under spinal anesthesia.

60 ASA I-III patients between 35-90 years of age who will be operated for femoral head/neck fractures will be included in the study. US-guided block procedure will be applied 30 minutes before the start of surgery. The patients will be divided into two groups, Group I, PENG block 20ml bupivacaine (n:30) and Group II, PENG block 30ml bupivacaine (n:30) using the closed envelope method in the operating room. Randomization will be performed by one of the researchers for each patient. Randomization information of patients will be used for all follow-up and data collection. The anesthetist applying the block will not take any part in collecting the data or performing the analysis. Numerical rating scale (NRS) will be used to evaluate pain. Patients will be given spinal anesthesia 30 minutes after PENG block. The primary outcome measure was determined as pain during positioning. NRS scores will be recorded after entering the operating room before, immediately before, during, and immediately after any analgesic intervention. Secondary outcome measures will be determined as the time required for LA performance (measured from the start of the position maneuvers to removal of the spinal needle), the quality of the patient position for LA performance ("unsatisfactory", "satisfactory", "good", "very good" to define SA). Questionnary 15 test will be applied to the patients 24 hours after the operation to measure patient satisfaction and to measure patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for total hip replacement surgery under spinal anesthesia
* ASA(American Society of Anesthesiology) 1-3
* Receiving consent that accept regional analgesia

Exclusion Criteria:

* contraindications for spinal anesthesia and PENG block
* impaired cognition or dementia
* multiple fractures

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Pain scores on the Numeric Rating Scale (NRS) | 30 minutes after intervention (PENG block) ]
  Changes in Numeric Rating Scale (NRS) at rest and on movement will be recorded at intervals. NRS is a unidimensional measure of pain intensity in adults. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

SECONDARY OUTCOMES:
Duration of spinal anesthesia performance | up to ten minutes
  It will be measured in "minutes", from the start of positioning maneuvers to the spinal needle removal
Quality of patient's position | up to ten minutes
  The position will be characterized as "unsatisfactory", "satisfactory", "good" or "very good"
analgesic consumption | 24 hours
  In the postoperative period, patients will be given opioids according to their pain density with a patient-controlled device, and the daily Morphine consumption in Patient Controlled Analgesia device will be collected and compared between groups.
Quality of recovery 15 scale | 24 hours after surgery
  Postoperative Quality of Recovery 15 in Turkish scale
Quadriceps weakness | postoperative 6th and 24th hours
  Quadriceps strength will be graded according to a 3-point scale: normal strength = 0 point (extension against resistance); paresis = 1 point (extension against gravity but not against resistance); and paralysis = 2 points (no extension).

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Ertas, specialist, Principal Investigator — samsun university, samsun training and research hospital
Locations (1):
- Samsun University, Samsun, Turkey (Türkiye)

REFERENCES:
- [Result] Zheng J, Pan D, Zheng B, Ruan X. Preoperative pericapsular nerve group (PENG) block for total hip arthroplasty: a randomized, placebo-controlled trial. Reg Anesth Pain Med. 2022 Mar;47(3):155-160. doi: 10.1136/rapm-2021-103228. Epub 2021 Dec 6. PMID 34873023